CLINICAL TRIAL: NCT03130036
Title: Biodistribution of [11C]Acetoacetate/[18F]Fluorodeoxyglucose in Subjects With Varying Risk Factors for Alzheimer's Disease and Subjects on a Diet Intervention
Brief Title: Biodistribution of [11C]Acetoacetate/[18F]Fluorodeoxyglucose in Subjects With Risk Factors for Alzheimer's Disease
Acronym: AcAc PET
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: IRB00033365
Record Dates: First submitted 2017-04-18; First posted 2017-04-26 (Actual); Last update posted 2025-07-28 (Actual); Status verified 2024-10

CONDITIONS: Mild Cognitive Impairment
Keywords: Memory; Cognitive
MeSH Terms: conditions — Cognitive Dysfunction

STUDY DESIGN:
Who Masked: Investigator
Masking Description: No masking is used
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- No risk of disease (Experimental): Subjects with no identifiable risk of Alzheimer's Disease
  Interventions: Other: [11C]Acetoacetate[18F]Fluorodeoxyglucose positron emission tomography scan
- Asymptomatic (Experimental): Asymptomatic subjects with increased risk of Alzheimer's disease
  Interventions: Other: [11C]Acetoacetate[18F]Fluorodeoxyglucose positron emission tomography scan
- Early Alzheimer's or Mild Cognitive Impairment (Experimental): Subjects with early Alzheimer's Disease or Mild Cognitive Impairment (MCI)
  Interventions: Other: [11C]Acetoacetate[18F]Fluorodeoxyglucose positron emission tomography scan

INTERVENTIONS:
Other: [11C]Acetoacetate[18F]Fluorodeoxyglucose positron emission tomography scan — A PET scan to measure uptake of acetoacetate and glucose in the brain will be administered to all participants enrolled in the study

SUMMARY:
This is a single center imaging study that will recruit 60 participants who are enrolled in the Effect of a Ketogenic Diet on Alzheimer's Disease Biomarkers and Symptoms: Brain Energy for Amyloid Transformation in AD (BEAT-AD) Study protocol. This cohort of patients will receive a maximum of 3 [11C]Acetoacetate (AcAc)/[18F]Fluorodeoxyglucose (FDG) PET scans over 18 weeks as part of this supplemental trial.

DETAILED DESCRIPTION:
The main objective of this study is to examine the brain biodistribution of [11C]AcAc/[18F]FDG, a proxy for acetoacetate (ketone body)/glucose metabolism in 3 study groups; 1) those without identifiable risk of Alzheimer's disease, 2) asymptomatic individuals with increased risk of Alzheimer's disease (such as pre diabetes),and 3) those with early Alzheimer's disease or MCI. Secondary objectives include determining the association between adipose tissue distribution/function and biomarkers of AD pathology.

ELIGIBILITY:
Inclusion Criteria:

* Mild cognitive impairment or subjective memory complaints
* Stable medical condition and medications
* Ability to complete baseline assessments

Exclusion Criteria:

* History of a clinically significant stroke
* Sensory impairment (visual, auditory)
* Diabetes requiring medication
* Current use of cholesterol/lipid lowering medications, anticonvulsants, drugs with potential interfering CNS effects (other than cholinesterase inhibitors or memantine), medications with significant anticholinergic activity, anti-parkinsonian medications or regular use of narcotic analgesics
* Untreated hypothyroidism or B12 deficiency

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2015-06-09 (Actual); Primary Completion 2024-06-19 (Actual); Study Completion 2024-06-19 (Actual)

PRIMARY OUTCOMES:
Brain biodistribution of [11C]AcAc | Baseline
  To assess brain metabolism of ketones (cerebral metabolic rate of acetoacetate/micromilliliters/100 g/min)
Brain biodistribution of [11C]AcAc | Change between baseline and four months
  To assess change in brain metabolism of ketones (cerebral metabolic rate of acetoacetate/micromilliliters/100 g/min)
Brain biodistribution of [18F]FDG - | Baseline
  To assess brain uptake of glucose (cerebral metabolic rate of glucose /micromilliliters/100 g/min)
Brain biodistribution of [18F]FDG - | Change between baseline and 4 months
  To assess change in brain uptake of glucose (cerebral metabolic rate of glucose /micromilliliters/100 g/min)

CONTACTS AND LOCATIONS:
Overall Officials: Suzanne Craft, PhD, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Wake Forest School of Medicine, Winston-Salem, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2023-12-19): https://cdn.clinicaltrials.gov/large-docs/36/NCT03130036/ICF_000.pdf